CLINICAL TRIAL: NCT05343520
Title: The Effect of Pelvic Floor Muscle Exercises Applied During Pregnancy on Genito-Pelvic Pain Level in Postpartum Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Husniye DINC KAYA, Associate Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 13022260-300-76447
Record Dates: First submitted 2022-03-17; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Genito-Pelvic Pain; Pelvic Floor Muscle Exercise; Pregnancy
Keywords: Pain; Exercise; Pregnancy; Genito-Pelvic; Postpartum
MeSH Terms: conditions — Pain; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The pregnant women who met the sampling criteria were assigned to the experimental or control groups with the numbers given by the generator on the website www.random.org. Odd numbers represented the experimental group, while even numbers represented the control group. In order to prevent the interaction of the pregnant women in the experimental and control groups with each other, a special examination room was arranged in the Antenatal Polyclinic and the study was carried out there. Pelvic floor muscle exercise was taught by the researcher (GY). Since the researcher knew which group the pregnant women in the sample were in, the study was single-blind. However, statistical analysis is double-blind because the statistics of the data are made by a different person.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): 30 pregnant women in the experimental group, pelvic floor muscle exercise was explained in detail and an exercise brochure was given in addition. Pelvic floor muscle exercises were taught by the researcher G.Y. In order for the exercise to be continued or applied correctly, the experimental group was interviewed by phone every 2 weeks. Information was given about continuing pelvic floor muscle exercises beginning from the 30th week of pregnancy until the postpartum 6th week.
  Interventions: Behavioral: Pelvic floor muscle exercises
- Control Group (No Intervention): The control group were filled only data collection forms

INTERVENTIONS:
Behavioral: Pelvic floor muscle exercises — Pelvic floor muscle exercises were applied to the pregnant women in the experimental group from the 30th gestational week to the 6th postpartum week.
  Arms: Experimental Group

SUMMARY:
Abstract Introduction and hypothesis The goal of the study is figuring out the effect of pelvic floor muscle exercises on genito-pelvic pain levels during the postpartum period.

Methods The data of the study, which was carried out in a randomized controlled experimental design, were collected in the antenatal policlinic of a public hospital between June-December 2019. There were 60 pregnant women in the experimental and control groups. Pelvic floor muscle exercises were applied to the pregnant women in the experimental group from the 30th week of gestation to the 6th postpartum week. The control group was not given pelvic floor muscle exercises training and only data collection forms were filled. During the study, the Descriptive Form, Verbal Category Scale, Pelvic Floor Distress Inventory-20, and Labour and Postpartum Information Form were applied to the pregnant women in both groups.

DETAILED DESCRIPTION:
Introduction Some important changes are observed on the pelvic floor musculature during the pregnancy and labour. Stretching occurs in nerve, muscle, fascia and ligament structures in the pelvic floor. This affects the pelvic floor musculature, causing dysfunction and pelvic pain. As a result of the study by Paterson et al. (2009), women stated that genito-pelvic pain started during pregnancy. Women reported that genito-pelvic pain was localized only on both sides of the genital area during pregnancy, and the pain was only in the genital area in the first days of the postpartum period.

It is estimated that genito-pelvic pain occurs in approximately 22% of pregnancy [3]. Acute genito-pelvic postpartum pain is a common problem regardless of vaginal delivery or caesarean section. Acute postpartum genito-pelvic pain rates can be up to 85%. This rate is observed as 92% one day after caesarean and vaginal delivery. Postpartum pain due to acute injuries from birth usually gets better in the first 2-3 months. However, for some new mothers, acute genito-pelvic pain may persist longer after delivery.

Considering that there are over 100 million births per year worldwide, the risk of women experiencing genito-pelvic pain increases accordingly. According to these estimations, at least one million women worldwide may suffer from persistent postpartum genito-pelvic pain for one year or more after giving birth. Acute genito-pelvic pain, on the other hand, negatively affects the recovery of the perineal region in the postpartum period, problems in bladder and bowel functions, and activities of daily living. Pelvic floor muscle exercises strengthen the pelvic floor muscles and increase urethral sphincter pressure. Strengthened pelvic floor muscles provide cushioning support to the pelvic organs and prevent pelvic organ prolapse and urinary incontinence by increasing urethral sphincter pressure (and promoting urethral muscle hypertrophy). They are also involved in sexual function and continence. Pelvic floor muscle exercises are exercises that provide the strength, endurance, contraction, relaxation or development of the pelvic floor muscles. In line with this literature, this study was conducted to determine the effect of pelvic floor muscle exercises applied during pregnancy on the level of genito-pelvic pain after delivery.

ELIGIBILITY:
Inclusion criteria for the study:

* Pregnant patients who want to join the study,
* Are primipara, not diagnosed with risky pregnancy,
* Are 30 weeks of gestation,
* Have no genito-pelvic pain pre-pregnancy,
* Have no vulvar varicosities,
* Are over the age of 18 and have no communication barrier (speaking Turkish)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant Women
Enrollment: 60 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
When the sample size was calculated using the G*Power Program with 95% power, 0.05 margin of error and 0.87 effect level, it was determined that at least 30 pregnant women should be recruited for each of the experimental and control groups. | Only 30th week of gestation
  Pelvic Floor Muscle Exercises effect measured with Descriptive Form
When the sample size was calculated using the G*Power Program with 95% power, 0.05 margin of error and 0.87 effect level, it was determined that at least 30 pregnant women should be recruited for each of the experimental and control groups. | 30th week of gestation
  Verbal Category Scale, The scale has 5 categories. It is cascaded from "Mild" to "Unbearable". Since it is a one-dimensional and verbal scale, it is very easy to apply. This scale is based on the patient choosing the most appropriate category to determine the level of pain. It is mostly preferred in acute pain or to measure the effect of the applied treatment. Although the application of the scale is simple, it also has disadvantages. The individual has to abide by the limited options in the questionnaire
When the sample size was calculated using the G*Power Program with 95% power, 0.05 margin of error and 0.87 effect level, it was determined that at least 30 pregnant women should be recruited for each of the experimental and control groups. | 6th postpartum week
  Verbal Category Scale, The scale has 5 categories. It is cascaded from "Mild" to "Unbearable". Since it is a one-dimensional and verbal scale, it is very easy to apply. This scale is based on the patient choosing the most appropriate category to determine the level of pain. It is mostly preferred in acute pain or to measure the effect of the applied treatment. Although the application of the scale is simple, it also has disadvantages. The individual has to abide by the limited options in the questionnaire
When the sample size was calculated using the G*Power Program with 95% power, 0.05 margin of error and 0.87 effect level, it was determined that at least 30 pregnant women should be recruited for each of the experimental and control groups. | 30th week of gestation
  Pelvic Floor Distress Inventory-20, The aim of the inventory created by Matthew D Barber et al. (2004) is to reveal the symptoms and level of all pelvic floor disorders seen in women. Its adaptation to Turkish and its validity-reliability were performed by physiotherapist Şeyda Toprak in 2010. The inventory consists of 3 sub-dimensions and contains 20 questions in total. The answer options for each question are divided into two as No and Yes. The Yes option is rated from "Insignificant" to "Very" in itself. No=0, and the level of the answer of Yes is Insignificant=1, Little=2, Moderate=3, Much=4 points. The number of points of the 3 sub-dimensions is summed up and a number between 0-300 points is obtained. The higher the score, the more serious the individual's problems are.
When the sample size was calculated using the G*Power Program with 95% power, 0.05 margin of error and 0.87 effect level, it was determined that at least 30 pregnant women should be recruited for each of the experimental and control groups. | 6th postpartum week
  Pelvic Floor Distress Inventory-20, The aim of the inventory created by Matthew D Barber et al. (2004) is to reveal the symptoms and level of all pelvic floor disorders seen in women. Its adaptation to Turkish and its validity-reliability were performed by physiotherapist Şeyda Toprak in 2010. The inventory consists of 3 sub-dimensions and contains 20 questions in total. The answer options for each question are divided into two as No and Yes. The Yes option is rated from "Insignificant" to "Very" in itself. No=0, and the level of the answer of Yes is Insignificant=1, Little=2, Moderate=3, Much=4 points. The number of points of the 3 sub-dimensions is summed up and a number between 0-300 points is obtained. The higher the score, the more serious the individual's problems are.
When the sample size was calculated using the G*Power Program with 95% power, 0.05 margin of error and 0.87 effect level, it was determined that at least 30 pregnant women should be recruited for each of the experimental and control groups. | Postpartum 72 nd hour
  Labour and Postpartum Information Form, A question form covering the 15 questions about the labour and postpartum problems.
When the sample size was calculated using the G*Power Program with 95% power, 0.05 margin of error and 0.87 effect level, it was determined that at least 30 pregnant women should be recruited for each of the experimental and control groups. | 6th postpartum week
  Labour and Postpartum Information Form, A question form covering the 15 questions about the labour and postpartum problems.

CONTACTS AND LOCATIONS:
Overall Officials: Husniye DINC KAYA, assoc.prof, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Gulcin Bozkurt, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Bortolini MA, Drutz HP, Lovatsis D, Alarab M. Vaginal delivery and pelvic floor dysfunction: current evidence and implications for future research. Int Urogynecol J. 2010 Aug;21(8):1025-30. doi: 10.1007/s00192-010-1146-9. Epub 2010 May 6. PMID 20445961
- [Background] Paterson LQ, Davis SN, Khalife S, Amsel R, Binik YM. Persistent genital and pelvic pain after childbirth. J Sex Med. 2009 Jan;6(1):215-21. doi: 10.1111/j.1743-6109.2008.01063.x. PMID 19170851
- [Background] Bartellas E, Crane JM, Daley M, Bennett KA, Hutchens D. Sexuality and sexual activity in pregnancy. BJOG. 2000 Aug;107(8):964-8. doi: 10.1111/j.1471-0528.2000.tb10397.x. PMID 10955426
- [Background] Vermelis JM, Wassen MM, Fiddelers AA, Nijhuis JG, Marcus MA. Prevalence and predictors of chronic pain after labor and delivery. Curr Opin Anaesthesiol. 2010 Jun;23(3):295-9. doi: 10.1097/aco.0b013e32833853e8. PMID 20446346
- [Background] Eisenach JC, Pan PH, Smiley R, Lavand'homme P, Landau R, Houle TT. Severity of acute pain after childbirth, but not type of delivery, predicts persistent pain and postpartum depression. Pain. 2008 Nov 15;140(1):87-94. doi: 10.1016/j.pain.2008.07.011. Epub 2008 Sep 24. PMID 18818022
- [Background] Declercq E, Cunningham DK, Johnson C, Sakala C. Mothers' reports of postpartum pain associated with vaginal and cesarean deliveries: results of a national survey. Birth. 2008 Mar;35(1):16-24. doi: 10.1111/j.1523-536X.2007.00207.x. PMID 18307483
- [Background] Rosen NO, Pukall C. Comparing the Prevalence, Risk Factors, and Repercussions of Postpartum Genito-Pelvic Pain and Dyspareunia. Sex Med Rev. 2016 Apr;4(2):126-135. doi: 10.1016/j.sxmr.2015.12.003. Epub 2016 Jan 11. PMID 27872022
- [Background] Thakar R, Stanton S. Management of genital prolapse. BMJ. 2002 May 25;324(7348):1258-62. doi: 10.1136/bmj.324.7348.1258. No abstract available. PMID 12028982
- [Background] Bo K, Frawley HC, Haylen BT, Abramov Y, Almeida FG, Berghmans B, Bortolini M, Dumoulin C, Gomes M, McClurg D, Meijlink J, Shelly E, Trabuco E, Walker C, Wells A. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for the conservative and nonpharmacological management of female pelvic floor dysfunction. Int Urogynecol J. 2017 Feb;28(2):191-213. doi: 10.1007/s00192-016-3123-4. Epub 2016 Dec 5. PMID 27921161
- [Derived] Yetiskin G, Dinc Kaya H. The effect of pelvic floor muscle exercises applied during pregnancy on genito-pelvic pain level in postpartum period. Int Urogynecol J. 2022 Oct;33(10):2791-2799. doi: 10.1007/s00192-022-05225-2. Epub 2022 Jun 9. PMID 35678835